CLINICAL TRIAL: NCT02742519
Title: A Phase 3b, 2-part, Randomized, Double-blind, Placebo-controlled Crossover Study With a Long-term Open-label Period to Investigate Ivacaftor in Subjects With Cystic Fibrosis Aged 3 Through 5 Years Who Have a Specified CFTR Gating Mutation
Brief Title: A Study to Evaluate Efficacy and Safety of Ivacaftor in Subjects With Cystic Fibrosis Aged 3 Through 5 Years Who Have a Specified CFTR Gating Mutation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VX15-770-123; 2015-001267-39 (EudraCT Number)
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part 1-Sequence 1 (Experimental): ivacaftor in Treatment Period 1 →washout→placebo in Treatment Period 2
  Interventions: Drug: ivacaftor; Drug: Placebo
- Part 1 - Sequence 2 (Experimental): placebo in Treatment Period 1→washout→ivacaftor in Treatment Period 2
  Interventions: Drug: ivacaftor; Drug: Placebo
- Part 2: ivacaftor (Experimental): open label period
  Interventions: Drug: ivacaftor

INTERVENTIONS:
Drug: ivacaftor
  Other Names: VX-770
Drug: Placebo
  Arms: Part 1 - Sequence 2; Part 1-Sequence 1

SUMMARY:
To evaluate the efficacy of ivacaftor treatment, as measured by lung clearance index (LCI), in subjects with cystic fibrosis (CF) who have a specified CF transmembrane conductance regulator (CFTR) gating mutation

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed diagnosis of CF.
* Must have 1 of the following CFTR gating mutations on at least 1 allele: G551D, G178R, S549N, S549R, G551S, G1244E, S1251N, S1255P, or G1349D.
* Hematology, serum chemistry, and coagulation at Screening with no clinically significant abnormalities or concomitant diagnosis that would interfere with the LCI and CT scan study assessments, as judged by the investigator.

Exclusion Criteria:

* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 4 weeks before Day 1
* Any clinically significant laboratory abnormalities at the Screening Visit that would interfere with the study assessments or pose an undue risk for the subject (in the opinion of the investigator)
* Abnormal liver function, at Screening, defined as ≥3 × upper limit of normal (ULN), of any 3 or more of the following: serum aspartate transaminase (AST), serum alanine transaminase (ALT), gamma-glutamyl transpeptidase (GGT), serum alkaline phosphatase (ALP), and total bilirubin
* History of solid organ or hematological transplantation
* Any clinically significant "non-CF-related" illness within 2 weeks before Day 1
* Use of any moderate or strong inducers or inhibitors of cytochrome P450 (CYP) 3A within 2 weeks before Day 1
* Participation in a clinical study involving administration of either an investigational or a marketed drug within 30 days or 5 terminal half-lives (whichever is longer or as determined by the local requirements) before Screening

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (4):
  - Parkville, Victoria
  - South Brisbane
  - Subiaco
  - Westmead
- Toronto, Ontario, Canada
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consisted of 2 parts: Part 1- Double Blind (DB) Crossover Treatment Period and Part 2- Open Label (OL) Period.
Groups:
- Part 1 Sequence 1: Ivacaftor First, Then Placebo: Ivacaftor administered every 12 hours for 8 weeks in treatment period 1 followed by placebo matched to Ivacaftor administered every 12 hours for 8 weeks in treatment period 2. Washout period of 8 weeks occurred between treatment period 1 and treatment period 2. For ivacaftor, the dose was either 50 milligram (mg) or 75 mg, as determined by the participant's body weight on Day 1.
- Part 1 Sequence 2: Placebo First, Then Ivacaftor: Placebo matched to Ivacaftor administered every 12 hours for 8 weeks in treatment period 1 followed by Ivacaftor administered every 12 hours for 8 weeks in treatment period 2. Washout period of 8 weeks occurred between treatment period 1 and treatment period 2. For ivacaftor, the dose was either 50 mg or 75 mg, as determined by the participant's body weight on Day 1.
- Part 2: Ivacaftor: Ivacaftor 50 mg, 75 mg or 150 mg, as determined by the participant's body weight at the beginning of Part 2, administered every 12 hours for up to 32 weeks in open label period.
Period: Part 1 Treatment Period 1 (8 Weeks)
Arm/Group | Part 1 Sequence 1: Ivacaftor First, Then Placebo | Part 1 Sequence 2: Placebo First, Then Ivacaftor | Part 2: Ivacaftor
Started | 8 | 6 | 0
Completed | 8 | 6 | 0
Not Completed | 0 | 0 | 0
Period: Part 1 Treatment Period 2 (8 Weeks)
Arm/Group | Part 1 Sequence 1: Ivacaftor First, Then Placebo | Part 1 Sequence 2: Placebo First, Then Ivacaftor | Part 2: Ivacaftor
Started | 8 | 6 | 0
Completed | 7 | 5 | 0
Not Completed | 1 | 1 | 0
Not completed — Availability of commercial drug | 1 | 1 | 0
Period: Part 2 Open Label Period (32 Weeks)
Arm/Group | Part 1 Sequence 1: Ivacaftor First, Then Placebo | Part 1 Sequence 2: Placebo First, Then Ivacaftor | Part 2: Ivacaftor
Started | 0 | 0 | 10 (Of 12 participants who completed DB period, only 10 entered OL period & 2 opted for commercial drug.)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 10
Not completed — Availability of commercial drug | 0 | 0 | 9
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Sequence 1: Ivacaftor First, Then Placebo | Part 1 Sequence 2: Placebo First, Then Ivacaftor | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.6 (0.7) | 4.2 (1.0) | 3.9 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Lung Clearance Index (LCI2.5) Through 8 Weeks of Treatment (Average of Week 4 and Week 8 LCI2.5)
Description: LCI2.5 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value.
Time Frame: Baseline Through Week 8 for each treatment period, Up to 24 Weeks
Population: Full Analysis Set (FAS) was used which included all randomized participants who had mutation on at least 1 allele, received at least 1 dose of study drug (Ivacaftor or placebo) and had at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Lung clearance index
Groups:
- Placebo (Crossover Part): Placebo matched to Ivacaftor administered orally every 12 hours for 8 weeks in treatment period 1 or treatment period 2.
- Ivacaftor (Crossover Part): Ivacaftor administered as determined by the participant's body weight on Day 1 orally every 12 hours for 8 weeks in treatment period 1 or treatment period 2.
Arm/Group | Placebo (Crossover Part) | Ivacaftor (Crossover Part)
Number analyzed (Participants) | 13 | 13
Lung clearance index | -0.07 (0.93) | -0.53 (1.23)
Statistical Analysis 1: Comparison: Placebo (Crossover Part) vs Ivacaftor (Crossover Part); Test type: Superiority; p = 0.2121, t-test, 2 sided

2. Secondary Outcome: Absolute Change From Baseline in Immunoreactive Trypsinogen Levels at Week 8
Description: Serum samples were collected for evaluation of change in immunoreactive trypsinogen levels at Week 8.
Time Frame: Baseline and Week 8 of each treatment period, Up to 24 Weeks
Population: FAS was used which included all randomized participants who had mutation on at least 1 allele, received at least 1 dose of study drug (Ivacaftor or placebo) and had at least 1 post-baseline assessment. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Placebo (Crossover Part) | Ivacaftor (Crossover Part)
Number analyzed (Participants) | 3 | 4
Nanogram per milliliter (ng/mL) | -9.3 (18.4) | -15.5 (6.5)

3. Secondary Outcome: Absolute Change From Baseline in Fecal Elastase-1 Levels at Week 8
Description: Fecal elastase-1 was used clinically to diagnose pancreatic exocrine insufficiency in participants with cystic fibrosis.
Time Frame: Baseline and Week 8 of each treatment period, Up to 24 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram per gram (mcg/g)
Arm/Group | Placebo (Crossover Part) | Ivacaftor (Crossover Part)
Number analyzed (Participants) | 11 | 10
microgram per gram (mcg/g) | -17.0 (55.4) | 23.1 (37.9)

4. Secondary Outcome: Absolute Change From Baseline in Weight at Week 8
Time Frame: Baseline and Week 8 of each treatment period, Up to 24 Weeks
Population: FAS was used which included all randomized participants who had mutation on at least 1 allele, received at least 1 dose of study drug (Ivacaftor or placebo) and had at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo (Crossover Part) | Ivacaftor (Crossover Part)
Number analyzed (Participants) | 13 | 13
Kilogram (kg) | 0.9 (1.0) | 1.1 (0.9)

5. Secondary Outcome: Absolute Change From Baseline in Body Mass Index (BMI) at Week 8
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).
Time Frame: Baseline and Week 8 of each treatment period, Up to 24 Weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilogram per meter square (kg/m^2)
Arm/Group | Placebo (Crossover Part) | Ivacaftor (Crossover Part)
Number analyzed (Participants) | 13 | 13
Kilogram per meter square (kg/m^2) | 0.13 (0.79) | 0.32 (0.59)

6. Secondary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to Month 15
Population: The Safety Set was used which included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Ivacaftor (Open Label Part): Ivacaftor administered as determined by the participant's body weight in the beginning of Part 2 orally every 12 hours in for up to 34 weeks in open label period.
Arm/Group | Placebo (Crossover Part) | Ivacaftor (Crossover Part) | Ivacaftor (Open Label Part)
Number analyzed (Participants) | 13 | 13 | 10
Participants
  Participants with any AEs | 11 | 11 | 6
  Participants with SAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Month 15
Groups:
- Ivacaftor (Crossover Part): Ivacaftor administered orally every 12 hours for 8 weeks in treatment period 1 or treatment period 2.
- Ivacaftor (Open Label Part): Ivacaftor administered orally every 12 hours in open label period.
Arm/Group | Placebo (Crossover Part) | Ivacaftor (Crossover Part) | Ivacaftor (Open Label Part)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 11/13 | 11/13 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Crossover Part) (N=13) | Ivacaftor (Crossover Part) (N=13) | Ivacaftor (Open Label Part) (N=10)
Haemophilus test positive (Investigations) | 0 | 1 | 1
Streptococcus test positive (Investigations) | 0 | 0 | 1
Bacterial test positive (Investigations) | 0 | 1 | 0
Pseudomonas test positive (Investigations) | 0 | 1 | 0
Cough (Skin and subcutaneous tissue disorders) | 3 | 2 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Bacterial disease carrier (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Vertex terminated the study early because of enrollment futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.

DOCUMENTS (2):
  • Study Protocol (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT02742519/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT02742519/SAP_001.pdf